CLINICAL TRIAL: NCT07392827
Title: Evaluation of the Effectiveness of Postoperative Pain Management in Pediatric Surgery Patients
Brief Title: Pediatric Postoperative Pain Management
Status: Active, not recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Nuriye Sidar ARSLAN, MD, Hacettepe University
Other Study IDs: SBA 25/704
Record Dates: First submitted 2026-01-27; First posted 2026-02-06 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Postoperative Pain; Pediatric Anesthesia Department; Regional Anaesthesia; Pain Scale; Caudal Epidural Anesthesia; Pediatric Surgical Patients
Keywords: Pediatric postoperative pain management
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 0-18 years old pediatric patiens: The main aim of this study is to evaluate all pediatric patients undergoing elective surgery; to accurately assess pain, the age groups were divided into 3. 0-59 months old patients will be evaluated with the FLACC scale, 60-84 months old patients' pain will be determined with the Wong-Baker FACES Scale, and 85 months-18 years old patients' pain will be assessed with the VAS score.

SUMMARY:
This prospective, observational study evaluates the effectiveness of perioperative pain management strategies in pediatric patients undergoing elective surgical procedures. Pediatric patients aged 0-18 years were assessed using age-appropriate pain scales during the first postoperative hour to measure acute pain control. Pain scores, emergence delirium evaluations, and interventions administered during routine clinical care were recorded to determine the effectiveness of standard pain management approaches across age and surgical subgroups. This study will not interfere with the clinician's treatment methods in any way. The treatments applied and their frequency will be determined. The success of the procedures performed will also be evaluated.

DETAILED DESCRIPTION:
Pain management in pediatric patients remains challenging despite advances in medical techniques. Limited availability of centers performing high-risk pediatric operations, narrow therapeutic dose ranges of medications used in children, and limited clinical experience contribute to persistent difficulties in pain management. Evidence indicates that many surgical patients experience acute postoperative pain, and a significant proportion do not receive adequate pain relief. Inadequate pain control has been associated with prolonged hospital stay, respiratory complications, infection, and delayed recovery.

Improvements in outcomes observed with advances in pain management techniques highlight the importance of effective postoperative analgesia in pediatric populations. Adequate pain control in the early postoperative period reduces complications and may prevent the development of chronic pain syndromes.

This prospective, observational study is designed to evaluate postoperative pain management strategies applied in pediatric patients undergoing elective surgical procedures performed by the Pediatric Surgery Department. The study focuses on the frequency and effectiveness of multimodal analgesia and regional anesthesia techniques used in routine clinical practice.

Pain management strategies in pediatric patients are supported by international pain societies; however, challenges persist due to concerns regarding invasive procedures in younger children, limitations in opioid use, and variability in clinical experience. Regional anesthesia techniques, neuraxial analgesia, and patient-controlled analgesia are routinely applied in the institution, and evaluation of their clinical effectiveness and complication rates is intended to contribute to existing literature.

The study is conducted in the Pediatric Surgery Operating Rooms of Hacettepe University Hospital and includes pediatric patients undergoing elective procedures under general anesthesia. Patients are stratified into age groups to account for differences in pain perception and assessment ability. Early postoperative evaluation includes assessment of recovery status to minimize the influence of postoperative delirium on pain scoring.

Postoperative pain assessment is performed using age-appropriate scales:

FLACC scale for children aged 0-5 years, Wong-Baker FACES scale for children aged 5-7 years, Visual Analog Scale (VAS) for children aged 7 years and older.

Data collection is performed prospectively. Following admission to the operating room, demographic characteristics, anesthesia techniques, surgical procedures performed, regional anesthesia applications, perioperative analgesic strategies, and intraoperative analgesic agents potentially affecting postoperative pain outcomes were recorded prospectively. Patients were monitored in the postoperative recovery unit for the first hour, which is considered the period during which acute postoperative pain is most intense. No modifications were made to routine anesthesia or analgesia practices, as the study was designed to observe and document routine clinical management without intervention.

Postoperative pain was assessed using age-appropriate scales. Pain scores ≥4 were considered indicative of pain requiring intervention, whereas scores ≥7 were accepted as reflecting insufficient pain control.

To differentiate pain-related agitation from postoperative emergence delirium, the Postoperative Anesthesia Emergence Delirium (PAED) scale was also used. Patients with PAED scores ≥10 were evaluated as having postoperative delirium. Because delirium may falsely elevate pain scores, pain assessments were performed concurrently with PAED evaluation after recovery. Pain assessment was repeated following the resolution of delirium symptoms. Patients whose delirium persisted despite appropriate treatment were excluded from analysis to prevent confounding effects on pain evaluation.

During the first postoperative hour, pain scores, PAED scores, and vital signs were recorded at 0 , 30, and 60 minutes in the recovery unit. Analgesic or delirium-related interventions administered according to clinical need, as well as the timing of these treatments, were also documented.

To improve comparability among procedures expected to produce similar postoperative pain levels, surgical interventions will be categorized into groups during data analysis. Pain outcomes and management strategies will be evaluated within comparable surgical and age subgroups to obtain a more homogeneous assessment of pain control success.Postoperative hospital stay duration is also recorded to evaluate potential associations between pain management success and recovery outcomes.

The study aims to provide observational data regarding current postoperative pain management practices pediatric surgical patients and to evaluate the effectiveness of routinely applied perioperative analgesic strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 0-18 years operated on by the Pediatric Surgery Department,
* Elective pediatric operations are performed under general anesthesia,
* ASA I-III group patients,

Exclusion Criteria:

* o Hemodynamically unstable patients. o ASA IV-VI group patients with life-threatening conditions. o Patients requiring emergency surgery.

  0 Patients requiring emergency surgery. o Patients over 18 years of age,
  * Patients admitted under sedation,
  * Non-surgical diagnostic or minimally invasive procedures such as gastroscopy, colonoscopy, bronchoscopy, and direct laryngoscopy,
  * Non-surgical needle biopsies,
  * Catheter placement and removal procedures,
  * Pain management interventions for chronic pain patients (TENS, Acupuncture),
  * Neurological (patients with chronic analgesic syndrome, peripheral neuropathies, spinal cord injury, cerebral palsy, meningomyelocele, multiple sclerosis, and neurodegenerative diseases) and mental developmental delay (autism spectrum disorders, mental retardation, Down syndrome),
  * Patients being followed up and treated for psychiatric illnesses (depression, anxiety disorder, somatization disorder, conversion disorder, schizophrenia, and bipolar disorder),
  * Patients with chronic pain syndrome or neuropathic pain who are using continuous analgesics in the preoperative period. Patients with a history of drug and psychoactive substance use, patients who are intubated postoperatively or monitored under intensive sedation for a long period, patients who are hemodynamically unstable in the postoperative period, patients who develop serious postoperative complications (hemorrhage, sepsis, MOOS), patients who require repeat surgery during the postoperative follow-up period, patients for whom Informed Consent could not be obtained will be excluded from the study.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Eligible pediatric patients undergoing elective surgery were consecutively enrolled during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-09-24 (Actual); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
0-59 months old age group pain intensity | Within the first postoperative hour (0, 30, and 60 minutes after recovery).
  Postoperative pain intensity was assessed using the FLACC (Face, Legs, Activity, Cry, Consolability) scale in pediatric patients aged 0-59 months. Pain scores ≥4 indicate moderate pain requiring intervention, whereas scores ≥7 indicate severe pain. Pain scores below 4 are defined as successful pain management.
  Score on FLACC scale (range 0-10)
60- 84 months old age group pain intensity | Within the first postoperative hour (0, 30, and 60 minutes after recovery).
  Postoperative pain intensity was assessed using the Wong-Baker FACES Pain Rating Scale in pediatric patients aged 60-84 months. Pain scores ≥4 indicate moderate pain requiring intervention, whereas scores ≥7 indicate severe pain. Pain scores below 4 are defined as successful pain management.
  Score on Wong-Baker FACES scale (range 0-10)
85 months -18 year of age group pain intensity | Within the first postoperative hour (0, 30, and 60 minutes after recovery).
  Postoperative pain assessed using the VAS (Visual Analog Scale) in patients aged 85 months-18 years. Scores ≥4 indicate pain requiring intervention; scores ≥7 indicate severe pain. Scores <4 indicate successful pain control.
  Unit of Measure:
  VAS score (0-10)

SECONDARY OUTCOMES:
Need for rescue analgesia in the postoperative recovery unit | Within the first postoperative hour (0, 30, and 60 minutes after recovery).
  Requirement for additional analgesic medication during the first postoperative hour in the recovery unit.
Postoperative emergence delirium assessed by the PAED scale | Within the first postoperative hour (0, 30, and 60 minutes after recovery).
  Emergence delirium assessed using the PAED (Pediatric Anesthesia Emergence Delirium) scale. Scores range from 0 to 20, with higher scores indicating more severe emergence delirium. A score of 10 or higher is considered consistent with postoperative emergence delirium. Delirium assessment is performed to avoid falsely elevated pain scores and to improve accuracy of postoperative pain evaluation. Patients whose PAED scores remain ≥10 during the first postoperative hour despite appropriate treatment are excluded from analysis.
  Unit of Measure:
  PAED score (0-20)

CONTACTS AND LOCATIONS:
Overall Officials: Filiz Uzumcugil, Professor Doctor, Study Director — Hacettepe University
Locations (1):
- Hacettepe University Hospital, Ankara, Altındag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided